CLINICAL TRIAL: NCT07385885
Title: Application of Ultrasound-guided Non-invasive Simulated Puncture Technique in Standardized Residency Training in Anesthesiology
Brief Title: Ultrasound-guided Non-invasive Simulation in Anesthesia Residency Training
Acronym: non-invasive
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hongwei Shi, Chief Physician, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20250922-KS-02
Record Dates: First submitted 2026-01-26; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Ultrasound; Needle; Residency; Anesthesiology; Training; Non-invasive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Method Teaching Group (No Intervention): Receive standardized theoretical instruction on ultrasound- guided peripheral nerve blocks; Be randomly assigned to conventional ultrasound scanning training;
- Non-invasive Simulated Puncture Teaching Group (Experimental): Receive standardized theoretical instruction on ultrasound- guided peripheral nerve blocks; Be randomly assigned to non-invasive simulated needle puncture training using an artificial intelligence-assisted system
  Interventions: Other: Non-invasive Simulated Puncture Teaching Group

INTERVENTIONS:
Other: Non-invasive Simulated Puncture Teaching Group — Receive standardized theoretical instruction on ultrasound- guided peripheral nerve blocks; Be randomly assigned to non-invasive simulated needle puncture training using an artificial intelligence-assisted system
  Arms: Non-invasive Simulated Puncture Teaching Group

SUMMARY:
Study Aim: This trial evaluates if a novel non-invasive, AI-assisted simulation training improves ultrasound-guided needle visualization skills in anesthesia residents.

Design: Trainees were randomized into two groups:

Intervention: AI-based, non-invasive simulated needle puncture training. Control: Conventional ultrasound teaching. Key Outcomes: The primary outcome is objective needle tip visibility. Secondary outcomes include anatomical identification, correct view acquisition, operator confidence, and overall scanning performance.

Assessment: Outcomes are measured via blinded expert evaluation and theoretical tests.

The goal of this randomized controlled clinical trial is to determine whether an ultrasound-guided non-invasive simulated needle puncture training technique can improve ultrasound-guided needle visualization skills in anesthesiology residents undergoing standardized residency training. The study is conducted in anesthesiology residents enrolled in a standardized residency training program.

The main questions it aims to answer are:

1. Does non-invasive simulated needle puncture training improve objective needle tip visibility during ultrasound-guided peripheral nerve block procedures?
2. Does this training method improve anatomical structure identification, acquisition of correct block views, operator confidence, and overall scanning performance compared with conventional ultrasound teaching? Researchers will compare a non-invasive simulated needle puncture training group with a conventional ultrasound teaching group to see if the simulated training technique leads to superior needle visualization and procedural performance.

Participants will:

Receive standardized theoretical instruction on ultrasound- guided peripheral nerve blocks; Be randomly assigned to either non-invasive simulated needle puncture training using an artificial intelligence-assisted system or conventional ultrasound scanning training; Perform ultrasound scanning and simulated or conventional practice on healthy volunteers; Undergo theoretical examinations and blinded expert assessments of ultrasound scanning performance and needle visualization outcomes.

DETAILED DESCRIPTION:
1. Teaching Implementation Prior to training, a questionnaire survey was used to collect basic information from the trainees. The course content was developed based on the following textbooks: Clinical Anesthesiology (4th Edition) edited by Guo Qulian and Yao Shanglong and published by People's Medical Publishing House; Modern Anesthesiology (4th Edition) edited by Deng Xiaoming et al. and published by People's Medical Publishing House; and Ultrasound-Guided Nerve Block Techniques edited by Wang Aizhong et al. and published by Shanghai Jiao Tong University Press.

   All participants initially attended a two-hour instructional course led by two teaching instructors. The course covered the techniques of interscalene brachial plexus, rectus sheath, adductor canal, and sciatic nerve blocks at the popliteal level. The content was based on the recent consensus project for basic ultrasound-guided blocks (Plan A) led by the British Association of Regional Anaesthesia, which defined strongly recommended structures for targeted scanning and block views. The specific structures included:

   Interscalene Brachial Plexus Block: Anterior scalene muscle; C5 nerve root; C6 nerve root; Middle scalene muscle.

   Rectus Sheath Block: Peritoneum; Rectus abdominis muscle; Anterior layer of the rectus sheath; Posterior layer of the rectus sheath.

   Adductor Canal Block: Femoral artery; Saphenous nerve; Sartorius muscle. Sciatic Nerve Block at the Popliteal Level: Common peroneal nerve; Tibial nerve. An additional structure, the popliteal artery, was also included in the block view for the popliteal sciatic nerve block.

   The teaching integrated practical case studies, images, videos, and other multimedia presentations. It focused on training ultrasound operation techniques, the acquisition of ultrasound images of nerves or tissue structures, structure identification, needle insertion methods, and puncture skills. This instruction aimed to establish a consistent scanning approach for each peripheral nerve block to minimize the influence of different scanning techniques on outcome measures.

   The instructional course also included familiarization with the Needle Trainer and the Sonosite Edge II ultrasound system, allowing participants to become acquainted with the equipment before evaluation. Two healthy volunteers (BMI 18.5-22 kg/m², aged 20-30 years) were recruited for ultrasound scanning practice.

   Participants in the experimental group used the Needle Trainer to perform non-invasive simulated puncture training for the four nerve blocks on healthy volunteers, utilizing a retractable virtual puncture needle. This training aimed to develop coordination between needle tracking and the ultrasound probe. Real-time ultrasound scanning provided color-highlighted displays of key ultrasound anatomical structures (the aforementioned four nerve blocks have CE/FDA certification). Participants in the control group used the Sonosite Edge II ultrasound system to perform scanning on healthy volunteers.

   Both groups prioritized hands-on practice, supplemented by instructor guidance. Participants were encouraged to ask questions at any time, with instructors providing real-time feedback, offering suggestions for improvement, and promptly adjusting participants' operation techniques and skills. Each participant received 12 minutes of ultrasound operation training per session. The training period spanned two weeks, followed by one week of clinical rotation. Both groups received equal training duration and identical instructional content.
2. Teaching Effectiveness Evaluation 2.1 Theoretical Assessment After the training, a theoretical examination was administered to participants from both groups. The exam focused on the identification of ultrasound anatomical structures and consisted of 25 multiple-choice questions. These questions were divided equally (5 questions each) into five sections: ultrasound basics and operation techniques, interscalene brachial plexus block, rectus sheath block, adductor canal block, and sciatic nerve block at the popliteal level. The total score was 100 points.

2.2 Practical Assessment A single expert, who was blinded to participant group allocation and had not been involved in the earlier instruction, assessed all participants. Each participant performed scans for the four nerve blocks on the same healthy volunteer. For each scan, timing (in seconds) began when the ultrasound probe touched the volunteer's skin and ended when the participant declared they had obtained the correct block view. At that moment, the ultrasound image was frozen and the time was recorded. The expert documented whether the obtained block view was correct (Yes/No). A correct block view was defined as one where the frozen image captured all structures identified during the earlier instruction.

Subsequently, the participant was asked to identify each strongly recommended structure for that specific peripheral nerve block on the original, unmodified ultrasound image displayed on the SonoSite machine. The expert recorded whether each structure identification was correct (Yes/No). Finally, for that scan, the expert gave the participant a global rating score for the scan on a scale from 0 (poor) to 10 (excellent).

For the clinical assessment (performing an adductor canal block on a patient), an experienced attending anesthesiologist or above was present to ensure patient safety and manage any emergent situations. The procedure was evaluated on-site by two experts in ultrasound-guided nerve blocks. The time taken for the nerve block procedure (from needle insertion to completion of the block) was recorded. All ultrasound imaging during each procedure was saved on the ultrasound machine's hard drive and transferred to a computer for subsequent analysis. The total procedure time was recorded from needle skin puncture until the needle tip was clearly visualized in the ultrasound image as successfully contacting the target. The number of puncture attempts was also recorded.

Upon completion of the procedure, the experts subjectively scored the visibility of the participant's needle tip on a scale from 1 (not visible) to 5 (very clear). An objective assessment of the dynamic images was performed using the method proposed by Hebard and Hocking [5]. All recorded ultrasound clips were reviewed independently by two blinded researchers using playback software. Clips were played back at slow speeds (1/4, 1/2 speed) and paused when necessary to precisely determine the presence or absence of the needle tip. The researchers measured the absolute time the needle tip was in view during each procedure (time visible) and calculated the percentage of time the needle tip was visible for each procedure (time visible / total procedure time × 100%), which we defined as the "objective needle tip visibility." The primary outcome measure was this needle tip visibility percentage.

Following this, the operator provided a confidence score regarding needle tip localization (1: no confidence at all, 2: slightly confident, 3: moderately confident, 4: quite confident, 5: very confident (able to accurately judge needle tip position)). Patient satisfaction with analgesia 30 minutes after the nerve block was assessed using an NRS score (0: extremely dissatisfied, 10: completely satisfied). The number of puncture attempts was recorded.

ELIGIBILITY:
Inclusion Criteria:

~Anesthesiology residents participating in the standardized residency training program in the Department of Anesthesiology at Nanjing First Hospital between October 2024 and October 2026.

Exclusion Criteria:

* Residents with prior experience in performing nerve block procedures.
* Residents currently participating in other teaching or research studies related to nerve blocks.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of needle tip visibility | After two weeks of training, followed by one week of clinical rotation
  For each procedure, investigators measured the absolute time during which the needle tip was visible on ultrasound (visible time) and calculated the percentage of needle tip visibility for each procedure (visible time / total procedure time × 100%), which was defined as objective needle tip visibility. The primary outcome measure of the study was the percentage of needle tip visibility.

SECONDARY OUTCOMES:
Accuracy of the acquired block view(s) | After two weeks of training, followed by one week of clinical rotation
  The expert assessed the correctness of block view acquisition (yes/no). A correct block view was defined as the presence of all predefined anatomical structures on the frozen ultrasound image.
Nerve block procedure time | procedure time
  Time from needle insertion to completion of the nerve block procedure
Number of needle insertion attempts | procedure time
  The number of puncture attempts was recorded
Expert-rated subjective needle tip visibility score | After two weeks of training, followed by one week of clinical rotation
  Expert(s) subjectively scored the needle tip visibility for each participant on a scale from 1 (invisible) to 5 (perfectly clear).
Time to obtain the correct block view | procedure time
  The time (in seconds) for each scan was measured from the moment the ultrasound probe made contact with the subject's skin until the participant declared that a correct block view had been obtained. At this point, the ultrasound image was frozen and the time was recorded.
Operator confidence score | After two weeks of training, followed by one week of clinical rotation
  The operator provided a confidence rating (1 = no confidence at all, 2 = slightly confident, 3 = moderately confident, 4 = quite confident, 5 = very confident (able to accurately identify the needle tip position)).
Expert global rating score of ultrasound scanning performance | After two weeks of training, followed by one week of clinical rotation
  The overall quality of each scan was rated by an expert on a 0-10 scale (0 = poor, 10 = excellent).

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Shi, Principal Investigator — Nanjing Hospital Affiliated to Nanjing Medical University
Locations (1):
- LiuHan, Nanjin, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Neal JM, Brull R, Horn JL, Liu SS, McCartney CJ, Perlas A, Salinas FV, Tsui BC. The Second American Society of Regional Anesthesia and Pain Medicine Evidence-Based Medicine Assessment of Ultrasound-Guided Regional Anesthesia: Executive Summary. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):181-94. doi: 10.1097/AAP.0000000000000331. PMID 26695878
- [Result] Soffler MI, Hayes MM, Smith CC. Central venous catheterization training: current perspectives on the role of simulation. Adv Med Educ Pract. 2018 May 25;9:395-403. doi: 10.2147/AMEP.S142605. eCollection 2018. PMID 29872360
- [Result] Chen XX, Trivedi V, AlSaflan AA, Todd SC, Tricco AC, McCartney CJL, Boet S. Ultrasound-Guided Regional Anesthesia Simulation Training: A Systematic Review. Reg Anesth Pain Med. 2017 Nov/Dec;42(6):741-750. doi: 10.1097/AAP.0000000000000639. PMID 28759501
- [Result] Bowness JS, Macfarlane AJR, Burckett-St Laurent D, Harris C, Margetts S, Morecroft M, Phillips D, Rees T, Sleep N, Vasalauskaite A, West S, Noble JA, Higham H. Evaluation of the impact of assistive artificial intelligence on ultrasound scanning for regional anaesthesia. Br J Anaesth. 2023 Feb;130(2):226-233. doi: 10.1016/j.bja.2022.07.049. Epub 2022 Sep 8. PMID 36088136
- [Result] Hebard S, Hocking G. Echogenic technology can improve needle visibility during ultrasound-guided regional anesthesia. Reg Anesth Pain Med. 2011 Mar-Apr;36(2):185-9. doi: 10.1097/aap.0b013e31820d4349. PMID 21425515
- [Result] Wiesmann T, Borntrager A, Zoremba M, Neff M, Wulf H, Steinfeldt T. Compound imaging technology and echogenic needle design: effects on needle visibility and tissue imaging. Reg Anesth Pain Med. 2013 Sep-Oct;38(5):452-5. doi: 10.1097/AAP.0b013e31829730d5. PMID 23759709